CLINICAL TRIAL: NCT01208597
Title: The Effectiveness of Adopting Humanized Service Program on Transvaginal Ultrasound About Women's Service Quality and Satisfaction.
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Ya-Ling Wu, Department of Obsterics and Gynecology
Other Study IDs: 99011
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Pregnant Women

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Owing to its image resolutions and its convenience in diagnosis, both better than abdominal ultrasound, transvaginal ultrasound is nowadays widely applied in diagnosing practice in obstetrics and gynecology. As a result, female examinees who undergo these check-up procedures have to expose their private parts, instead of their abdomens like the old days. According to the literature, women who receive transvaginal ultrasound check-ups normally have anxiety reactions, and worry about pain and discomfort. In clinical practice, when giving advice to the examinees to go through this check-up, more than often the diagnosis itself is its sole purpose, and little psychological assistance is offered. Traditional clinical space and disposal process tend to be designed to serve the purposes of conforming to the customs of medical staff and to the integrity of human resources and facilities in the hospital managers' minds, and less frequently tend to take the needs of patients into consideration. Consequently these patients are forced to enter strange medical environments and accommodate to the existent medical systems, with physical and psychological discomforts, to suffer from even more uncomfortable and anxiety-causing check-ups. Current medical service is required to not only provide a clean environment, but also give attention to creating an artistic space to increase healthy factors to the environment. The literature points out that a comfortable and artistic space can eliminate environmental strangeness, and help patients to soothe their pressures caused by their own and by the environment.

DETAILED DESCRIPTION:
This women-centered study designs a "humanized service program", to give women care and respect, and protect women's privacy and their rights to know; the space design is women-concerned, warm and homelike-layout; its furnishings are well-designed in order to facilitate access for women to use, and give every effort to maintain women's safety, comfort and self-esteem. The main purpose of this space is to provide the women who receive transvaginal ultrasound "the human-based check-up service program", in order to see how it affects the physical and psychological experiences of these women, its service quality and service satisfaction.

This study adopts a quasi-experimental research method and takes the ultrasound examination rooms of the obstetrics and gynecology department of a medical center in northern Taiwan as the sites of collecting case data. The studied targets are the women who came to the obstetrics and gynecology clinic as outpatients and were required to undergo transvaginal ultrasound. The women in the control-group were offered with "the routine service", and the experimental group, the "humanized service program". The study results compare differences between the control group and the experimental group with regard to their respective basic information concerning their physical and psychological experiences, their opinions on its service quality and service satisfaction, discuss about the effectiveness of this program, and explore the inter-relationships among the physical and psychological experiences, service quality and service satisfaction. The research tools include the humanized service programs and the research questionnaires. The research questionnaires include a basic information scale, a physical and psychological experiences scale, a service quality scale and a service satisfaction scale. Scales of humanized service programs and basic information adopt expert validity for validity evaluation; the physical and psychological experiences scale, the service quality scale and the service satisfaction scale adopt expert validity and internal consistency reliability and construct validity for reliability and validity evaluation. The results show that its reliability and validity both fall within acceptable ranges.

Chi-square test analysis reveals that the cases in the two groups have homogeneity. From the descriptive statistics, it can be learned that the 9 most common existing feelings the women had who received transvaginal ultrasound are the following: sense of tension over the whole body, feeling nervous, feeling awkward , feeling shy, feeling embarrassed, worrying about discomfort, worrying about pain, fear of infection and lower abdominal fullness feeling. The outpatients in the two groups perceived the service quality dimensions as such: the highest dimension is the Empathy, and the lowest is the Tangibles. The highest dimension of the two groups concerning the check-up service satisfaction is the Staff's Attitude, and the lowest is the environment and the Waiting Time for Check-Up. Independent-samples T test analysis shows that the points of the cases in the experimental group are significantly higher than the ones of the control group in these three aspects: physical and psychological experience, service quality and service satisfaction. This study results demonstrates that the human-based check-up service program is effective for physical and psychological experiences, service qualities and satisfaction. It lessens the physical and psychological negative feelings of the women when they underwent transvaginal ultrasound, and at the same time improves the transvaginal ultrasound service quality and satisfaction. Structural Equation Modeling (SEM) analysis of the relationships among the three, physical and psychological experience, service quality and service satisfaction, shows that there is a significant positive correlation between service quality and physical and psychological experiences, also between service quality and service satisfaction. Moreover, the service quality produces an indirect effect on service satisfaction through the physical and psychological experience. There is also a significant positive correlation between physical and mental feelings and service satisfaction; this indicates that increase in service quality may affect the physical and psychological experience of women to tend to be positive, and enlarge service satisfaction; when women have more positive physical and mental feelings, it will also increase their satisfaction with the services.

The physical and psychological experience scale designed in this study can be applied to other assessments of women's physical and psychological feelings under the situations of necessary perineal area exposures, such as Pap smear, colposcopy and so on. "The humanized service program" can offer the transvaginal ultrasound examinees better service; besides, it can be used in various female-based obstetrics and gynecology-related check-ups. Within other medical divisions, this concept can also be applied in order to provide more superior medical service and care.

ELIGIBILITY:
Inclusion Criteria:

1. More than 20 years of sexual experience in adult women.
2. Clear consciousness, those without severe cognitive impairment, such as dementia, mental retardation or mental illness.
3. Literacy and the use of Chinese or Taiwanese.
4. Willingness to participate in the research.

Exclusion Criteria:

1. virgin
2. Refused to participate in the research

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult women
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-02; Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Ling Wu, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University WanFang Hospital, Taipei, Taiwan